CLINICAL TRIAL: NCT00170911
Title: Efficacy and Safety of AAE581 in Postmenopausal Women With Osteopenia/Osteoporosis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE581A1201
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Postmenopausal women; Cathepsin K inhibitor
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: AAE581

SUMMARY:
AAE581 is a specific inhibitor of the cysteine protease cathepsin K. This trial is designed to provide detailed information about the effects( efficacy and safety) of AAE581 on Bone Mineral Density.

ELIGIBILITY:
Inclusion Criteria:

* Low spine Bone Mineral Density
* 0 to 1 prevalent fracture in non lumber spine

Exclusion Criteria:

* History or presence of any bone disease other than osteopenia /osteoporosis
* Previous treatment with other anti-osteoporosis agent(Wash out required)
* Evidence of vitamin D deficiency

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 50 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-03; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change of lumbar spine(L1-L4)BMD at 12 months
Safety of 12 month treatment

SECONDARY OUTCOMES:
Change of BMD of lumbar spine(L1-L4,L2-L4)、total hip, femoral neck, forearm and total body at 3, 6, 9 and 12 months
Change of Bone markers(Serum CTX,P1NP, OC, BSAP and urinary NTX, DPyr at 1,3,6,9 and 12 months
Plasma concentration of AAE581 and AEE325 at 1,3,6,9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Sponsor GmbH